CLINICAL TRIAL: NCT04442958
Title: Effectiveness of Convalescent Immune Plasma Therapy in Severe COVID-19 Patients With Acute Respiratory Distress Syndrome
Brief Title: Effectiveness of Convalescent Immune Plasma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020.05.2.14.070
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convalescent Plasma Therapy Group (Experimental): One dose of 200 mL of convalescent ımmune plasma derived from recently recovered donors with the neutralizing antibody titers above 1:640 was transfused to the patients as an addition to standart critical care treatment.
  Interventions: Other: Convalescent Immune Plasma
- Non-Plasma Therapy Group (No Intervention): Standart critical care treatment group

INTERVENTIONS:
Other: Convalescent Immune Plasma — One dose of 200 mL of convalescent ımmune plasma derived from recently recovered donors with the neutralizing antibody titers above 1:640 was transfused to the patients as an addition to standart critical care treatment.
  Arms: Convalescent Plasma Therapy Group

SUMMARY:
The aim of the study is to evaluate the safety, improvement of clinical symptoms and laboratory parameters of convalescent immune plasma treatment in severe Covid-19 patients with ARDS.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the safety, improvement of clinical symptoms with hypoxemia, metabolic and laboratory parameters of patients with convalescent immune plasma treatment in severe Covid-19 patients followed up in critical care unit.

ELIGIBILITY:
Inclusion Criteria Clinical diagnosis of Covid-19

Exclusion Criteria Age lower than 18 Lower plasma IgA levels PaO2/FiO2 higher than 300 mmHg SpO2 higher than 90

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Plasma ferritin level | 7. day
  Acute phase reactant
Lymphocyte count | 7. day
  Infection markers
D-Dimer level | 7. day
  Hypercoagulability
C-Reactive protein level | 7. day
  Infection markers
Plasma procalcitonin level | 7. day
  Infection markers
Plasma fibrinogen level | 7. day
  Coagulopathy

SECONDARY OUTCOMES:
Fractional Inspired Oxygen Level | 7. day
  Arterial oxygenation
Partial Oxygen Saturation level | 7. day
  Arterial oxygenation
Arterial Oxygen level | 7. day
  Arterial oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Salih SS Sevdi, Md, Principal Investigator — Istanbul Bagcılar Training and Research Hospital
Locations (1):
- Istanbul Bagcılar Training and Research Hospital, Istanbul, Turkey (Türkiye)